CLINICAL TRIAL: NCT02770833
Title: Acute Effects of Different Protein Sources and Different Glycemic Index on Energy Balance, Glucose Allostasis and Amino Acid Metabolism.
Brief Title: Acute Effects of Different Protein Sources and Different Glycemic Index on Energy Balance, Glucose Allostasis and Amino Acid Metabolism: a Randomized, 4-condition, Two Cross-over Study in Adults.
Acronym: FINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Fisheries and Aquaculture Industry Research Fund (Other); National Institute of Nutrition and Seafood Research, Norway (Other Government)
Responsible Party: Principal Investigator, Anne Birgitte Raben, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H-1-2014-038 (B314)
Record Dates: First submitted 2014-10-29; First posted 2016-05-12 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Overweight
Keywords: Proteins (seafood and meat); GI; Energy expenditure; Energy balance; Thermogenesis (DIT); Appetite regulating hormones; Appetite sensations; Glucose allostatis; Amino acid metabolism; Satiety; Food preferences
MeSH Terms: conditions — Overweight; Food Preferences | interventions — In Situ Hybridization, Fluorescence; Red Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salmon vs. veal and CHO with low or high GI (Experimental): In the first clinical study (Study 1), subjects will eat salmon or veal combined with high or low GI carbohydrates. Each subject will be engaged in each of the following four 1-day test meals:
  * Meat balls with salmon served with tomato sauce and other accompaniments with low GI
  * Meat balls with salmon served with tomato sauce and other accompaniments with high GI
  * Meat balls with veal served with tomato sauce and other accompaniments with low GI
  * Meat balls with veal served with tomato sauce and other accompaniments with high GI
  Interventions: Other: Fish and carbohydrats with low or high GI; Other: Veal and carbohydrats with low or high GI
- Cod vs. veal and CHO with low or high GI (Experimental): In the second clinical study (Study 2), subjects will eat codfish or veal combined with high or low GI carbohydrates. Each subject will be engaged in each of the following four 1-day test meals:
  * Meat balls with codfish served with tomato sauce and other accompaniments with low GI
  * Meat balls with codfish served with tomato sauce and other accompaniments with high GI
  * Meat balls with veal served with tomato sauce and other accompaniments with low GI
  * Meat balls with veal served with tomato sauce and other accompaniments with high GI
  Interventions: Other: Fish and carbohydrats with low or high GI; Other: Veal and carbohydrats with low or high GI

INTERVENTIONS:
Other: Fish and carbohydrats with low or high GI
Other: Veal and carbohydrats with low or high GI

SUMMARY:
The hypothesis is that seafood proteins given in combination with carbohydrates with low GI are superior to seafood proteins in combination with carbohydrates with high GI and meat in combination with both carbohydrates with low and high GI in promoting energy expenditure and satiety. The overall objective of this study is to investigate the acute effects of meals containing fish versus meat proteins on energy balance (thermogenesis, appetite regulating hormones and appetite sensations), markers of glucose allostatis and amino acid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Between 18 and 50 years of age
* BMI between 25.0 and 30.0 kg×m-2
* Fasting blood glucose < 5.9 mmol/L (measured at the screenings visit)
* Non-smoker

Exclusion Criteria:

* Self-reported eating disorders or irregular eating schedule (e.g. skipping breakfast)
* Chronic diseases (e.g. cancer, asthma, back pain, thyroid disease, heart disease, diabetes, neurological disorders, or sleep disorders)
* Use currently or within the previous 3 months of prescription medication that has the potential of affecting body weight or glucose metabolism such as glucocorticoids (but excluding inhaled and topical steroids; bronchodilators are allowed), psychoactive medication, epileptic medication, or weight loss medications (either prescription, over the counter or herbal). Low dose antidepressants are allowed if they, in the judgement of the investigator, do not affect weight or participation to the study protocol. Levothyroxine for treatment of hypothyroidism is allowed if the participant has been on a stable dose for at least 3 months.
* Women who are pregnant, breast-feeding or have intention of becoming pregnant during the study period
* Menopausal women and women with an irregular menstrual cycle
* Food allergies
* Substance abuse
* Vigorous physical activity more than 10 hours/week
* Alcohol intake above the recommendations from the Danish Health and Medicines Authority
* Caffeine intake above 300 mg/day
* Night- or shift work
* Blood donation <1 month before study commencement and during study period
* Simultaneous participation in other clinical studies
* Inability, physically or mentally, to comply with the procedures required by the study protocol, as evaluated by the study staff
* Subject's general condition contraindicates continuing the study, as judged by the study personnel or the medical expert

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Differences in diet induced thermogenesis between the four test meals | 3 hours
  In the following three hours after eating the test meal respiratory gas exchange will be measured 6x25 minutes with 5 minutes breaks in between each measurement. Diet induced thermogenesis (DIT) will be measured by indirect calorimetry using a ventilated hood system. Each measurement will last for 25 minutes of which the last 20 minutes will be used for calculation of energy expenditure.

SECONDARY OUTCOMES:
Satiety | 3 hours
  Evaluated by VAS-measures of subjective appetite sensations (satiety, hunger, fullness and prospective food consumption)
Food preferences | 3 hours
  In an attempt to measure spontaneous energy intake and macronutrient preferences in an experimental context, the participants will be given an ad libitum buffet lunch at noon. A cold and hot buffet-style lunch comprising a variety of foods (representing a wide selection of food groups) will be offered after the last measurement of gas exchange and the participants will be instructed to eat ad libitum.
Glucose | 3 hours
  Blood sample
Insulin | 3 hours
  Blood sample
Glucagon | 3 hours
  Blood sample
C-peptide | 3 hours
  Blood sample
Plasma amino acids | 3 hours
  Blood samples
Appetite regulating hormones | 3 hours
  e.g. glucagon-like peptide-1 (GLP-1)
Free fatty acids | 3 hours
  Blood sample
Glycerol | 3 hours
  Blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Anne Raben, Prof, Principal Investigator — Prof at the department of Nutrition, Exercise and Sports
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Frederiksberg, Denmark